CLINICAL TRIAL: NCT06034964
Title: Retrospective Study of Tislelizumab Combined With Chemotherapy in First-line Treatment of HER2-negative Advanced Gastric Cancer
Brief Title: Tislelizumab Combined With Chemotherapy in First-line Treatment of AGC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: NCC3221
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Tislelizumab; Chemotherapy; First-line; Gastric Cancer Stage IV
Keywords: Tislelizumab; First-line; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab：200mg, iv, d1, 21 days per cycle, until disease progression or intolerable toxicity
  Other Names: BGB-A317

SUMMARY:
This is a single-center, retrospective clinical study to evaluate the efficacy and safety of tislelizumab combined with first-line chemotherapy in the treatment of HER2-negative advanced gastric cancer.

DETAILED DESCRIPTION:
This study aims to include 60 HER-2 negative advanced gastric cancer patients who received first-line treatment with tislelizumab combined with chemotherapy in our hospital from November 1, 2020 to November 1, 2021. Clinicopathological data, blood tests and imaging data of the patients were collected. The primary endpoints evaluated were PFS and OS, and the secondary endpoints were ORR and safety. At the same time, ctDNA and peripheral cytokine status of patients as well as second-generation sequencing of tumor tissues at baseline were collected for the exploration of therapeutic efficacy related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with initially unresectable (locally advanced or metastatic) or postoperative recurrence of gastric adenocarcinoma or gastroesophageal junction adenocarcinoma confirmed by histopathology have not received any anti-tumor treatment for advanced gastric cancer in the past;
2. Pathological immunohistochemistry or FISH detection of gastric cancer tissue indicates negative Her-2;
3. Age range from 18 to 70 years old, regardless of gender;
4. The distance between postoperative recurrence and the end of neoadjuvant/adjuvant chemotherapy is more than 6 months;
5. If the patient experiences toxic side effects after receiving new adjuvant/adjuvant treatment, they need to recover from previous treatment toxic side effects to ≤ 1 level; According to the RECIST evaluation criteria, there should be at least one assessable lesion. Expected survival time ≥ 3 months;

7. ECOG score ≤ 2 points; 8. Main organ functions are basically normal, blood count (within 7 days): hemoglobin ≥ 90g/L, white blood cells ≥ 4.0 × 109/L, neutrophils ≥ 2.0 × 109/L, platelet ≥ 100.0 × 109/L. Total bilirubin 1.0 UNL, creatinine 1.0 × UNL, AST/ALT 2.5 UNL. Liver metastasis: ASAT/ALAT 5 UNL; 9. The electrocardiogram/cardiac function tests are basically normal.

Exclusion Criteria:

1. Suffering from undifferentiated gastric cancer or squamous cell carcinoma of the gastroesophageal junction and other pathological types of malignant tumors;
2. Have received anti-tumor treatment for gastric adenocarcinoma or adenocarcinoma at the junction of stomach and esophagus that can not be operated on for the first time or recur after operation, including but not limited to chemotherapy, Targeted therapy, immunotherapy, etc. (except for Thymosin and traditional Chinese medicine treatment);
3. Patients with other primary malignant tumors other than gastric cancer, excluding cured skin Basal-cell carcinoma and cervical Carcinoma in situ;
4. Patients with simple or combined brain metastasis;
5. Has experienced gastrointestinal perforation or fistula within 6 months prior to enrollment;
6. Patients who also suffer from other important organ diseases, including severe heart disease;
7. Complications such as uncontrollable moderate to massive ascites, active gastrointestinal bleeding, gastrointestinal perforation, gastrointestinal obstruction, etc;
8. Patients with chronic diseases such as hypertension, hyperglycemia, and COPD that are difficult to control;
9. Those who require antibiotics for systemic anti infection, active hepatitis, active pulmonary tuberculosis, and other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER-2 negative, untreated patients with advanced gastric cancer.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression-free Survival
OS | 3 years
  Overall Survival

SECONDARY OUTCOMES:
ORR | 2 years
  Objective Remission Rate
DCR | 2 years
  Disease Control Rate
DOR | 2 years
  Duration of Remission
Safety and Tolerability | 2 years
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yang, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China